CLINICAL TRIAL: NCT03118505
Title: A Prospective, Randomized, Multi-Center, Open-Label Pilot Study of Infuse® Bone Graft With Mastergraft® Strip and Posterior Fixation for Posterolateral Fusion (PLF) Treatment of Multi-Level Degenerative Lumbosacral Spinal Conditions
Brief Title: A Study of Infuse® Bone Graft With Mastergraft® Strip and Posterior Fixation for Posterolateral Fusion (PLF) Treatment of Multi-Level Degenerative Lumbosacral Spinal Conditions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P16-03
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Multi-Level Degenerative Lumbosacral Spinal Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Group 1 (Experimental): Infuse Bone Graft [4.2 mg per operative level] + Mastergraft Strip + local bone autograft + posterior fixation
  Interventions: Device: Infuse Bone Graft
- Group 2 (Experimental): Infuse Bone Graft [6 mg per operative level] + Mastergraft Strip + local bone autograft + posterior fixation
  Interventions: Device: Infuse Bone Graft
- Group 3 (Experimental): Infuse Bone Graft [12 mg per operative level] + Mastergraft Strip + local bone autograft + posterior fixation
  Interventions: Device: Infuse Bone Graft
- Control (Active Comparator): Medtronic DBM + local bone autograft (and supplemented with iliac crest bone graft (ICBG), if needed) + posterior fixation.
  Interventions: Device: Medtronic DBM

INTERVENTIONS:
Device: Infuse Bone Graft — Infuse Bone Graft + Mastergraft Strip + local bone autograft + posterior fixation
  Arms: Group 1; Group 2; Group 3
Device: Medtronic DBM — Medtronic DBM + local bone autograft (and supplemented with iliac crest bone graft (ICBG), if needed) + posterior fixation
  Arms: Control

SUMMARY:
The purpose of this study is to obtain safety and effectiveness data on the investigational device for multi-level PLF procedures and determine the most appropriate rhBMP-2 dose for use in this indication. The study information may be used for a potential pivotal study design.

ELIGIBILITY:
Inclusion Criteria:

1. Degenerative lumbar spine condition:

   1. Requiring a PLF procedure using a bilateral metallic screw and rod system in 2-4 consecutive levels from L2-S1; and
   2. Diagnosed with: instability (up to and including Grade 2 spondylolisthesis, retrolisthesis, or lateral listhesis), stenosis with documented pre-operative instability, and/or recurrent disc herniation, any of which may have possible concomitant lumbar degenerative deformity (Cobb angle ≤ 30 degrees).
2. Preoperative ODI score ≥40.
3. Preoperative pain score of ≥8 (out of 20) on the Preoperative Leg Pain Questionnaire.
4. Most inferior treated spinal level is able to accommodate an interbody fusion device.
5. ≥21 years of age at the time of signing the informed consent.
6. Failed ≥6 months non-operative treatment (e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS).
7. Is willing and able to comply with the study plan and able to understand and sign the Subject Informed Consent Form.

Exclusion Criteria:

1. Prior spinal fusion surgical procedure at the involved or adjacent spinal levels. (Prior non-fusion surgery at the target levels, including discectomy and/or single-level foraminotomy or laminectomy, is allowed.)
2. Prior lumbar disc arthroplasty.
3. Significant lumbar instability, defined as sagittal listhesis >Grade 2 at any involved level using Meyerding's Classification or lateral listhesis >25% lateral translation at any involved level.
4. Planned use of an internal or external bone growth stimulator.
5. Lumbar scoliosis >30 degrees.
6. Osteoporosis to a degree that spinal instrumentation is contraindicated or a history of atraumatic vertebral fracture.
7. Morbidly obese, as defined by a Body Mass Index (BMI) >40.
8. Presence of active malignancy or prior history of malignancy.
9. Overt or active bacterial infection, either local or systemic.
10. Has undergone systemic administration of any type of corticosteroid, anti-neoplastic, immunostimulating, or immunosuppressive agents within 30 days prior to implantation of the assigned treatment.
11. Comorbidities precluding subject from being a surgical candidate.
12. History of autoimmune disease known to affect bone metabolism or the spine (e.g., spondyloarthropathies, juvenile arthritis, rheumatoid arthritis, Graves' disease, Hashimoto's thyroiditis).
13. History of any endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta).
14. History of exposure to any recombinant proteins used for bone formation (i.e., Infuse Bone Graft, OP-1 Putty, OP-1 Implant, AUGMENT Bone Graft, GEM21S, i-FACTOR Peptide Enhanced Bone Graft, or PepGen P-15 Synthetic Bone Graft).
15. Hypersensitivity or allergy to any components of the study treatments including, but not limited to, bone morphogenetic proteins (BMPs); injectable collagen; protein pharmaceuticals (e.g., monoclonal antibodies or gamma globulins); bovine collagen products; gentamicin or glycerol (which may be present in trace amounts in the DBM products); and/or instrumentation materials (titanium, titanium alloy, cobalt chrome, cobalt chrome alloy, or polyetheretherketone [PEEK]).
16. History of any allergy resulting in anaphylaxis.
17. Is a prisoner.
18. Is mentally incompetent. If questionable, obtain psychiatric consult.
19. Treatment with an investigational therapy (drug, device, and/or biologic) within 30 days prior to implantation surgery, or such treatment is planned during the 24-month period following implantation of the study treatment.
20. Pregnant or nursing. Females of child-bearing potential must agree not to become pregnant for one year following surgery.
21. Any condition that would interfere with the subject's ability to comply with study instructions, might confound the interpretation of the study, or put the subject at risk.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-29 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radiological Fusion Success | 12 months
  Fusion at each treated level is defined as radiological fusion assessed by radiograph and CT. A subject will be considered a fusion success when the following criteria are met for each treated level:
  * Bilateral bridging bone (superior transverse process to the inferior transverse process) at each treated level (CT);
  * No more than 3mm translational motion and less than 5 degrees in angular motion at each treated level (flexion/extension radiographs); and
  * Absence of cracking, as evidenced by radiolucent lines completely through the fusion mass (all radiograph views).

SECONDARY OUTCOMES:
Overall success rate at 12 and 24 months | 12 and 24 months
  Overall success is defined as the participant who meet the following five criteria:
  * Radiographic success, defined as radiological fusion success in the posterolateral space;
  * Pain/disability (ODI) success, defined as at least a 15-point improvement from baseline;
  * Neurological success, defined as maintenance or improvement in neurological status;
  * No SAE related to the PLF grafting material or posterior fixation; and
  * No secondary surgeries classified as a "failure."
ODI score at 12 and 24 months | 12 and 24 months
  The self-administered Oswestry Disability Index (ODI) Questionnaire (Version 2.1) will be used to assess patient pain and ability to function. The ODI scale ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
ODI success rate at 12 and 24 months | 12 and 24 months
  ODI success is defined as at least a 15-point improvement from baseline.
Neurological success rate at 12 and 24 months | 12 and 24 months
  Overall neurological success is defined as maintenance or improvement in four key neurological assessments: motor function, sensory function, reflexes, and straight leg raise. In order to be considered a success, each element in the motor, sensory, reflexes, and straight leg raise examinations must remain the same or improve from the time of the preoperative evaluation to the time period evaluated.
Back pain score at 12 and 24 months | 12 and 24 months
  Numerical rating scales, adapted in part from Measuring Health, will be used to evaluate back pain. The back pain score (0-20) is the summation of pain intensity (0-10) and duration (0-10) scores.
Back pain success at 12 and 24 months | 12 and 24 months
  Back pain success is defined as at least 30% improvement from baseline.
Leg pain score at 12 and 24 months | 12 and 24 months
  Numerical rating scales, adapted in part from Measuring Health, will be used to evaluate leg pain. The leg pain score (0-20) is the summation of pain intensity (0-10) and duration (0-10) scores.
Leg pain success at 12 and 24 months | 12 and 24 months
  Leg pain success is defined as at least 30% improvement from baseline.
Radiological fusion success rate at 24 months | 24 months
  Fusion at each treated level is defined as radiological fusion assessed by radiograph and CT. A subject will be considered a fusion success when the following criteria are met for each treated level:
  * Bilateral bridging bone (superior transverse process to the inferior transverse process) at each treated level (CT);
  * No more than 3mm translational motion and less than 5 degrees in angular motion at each treated level (flexion/extension radiographs); and
  * Absence of cracking, as evidenced by radiolucent lines completely through the fusion mass (all radiograph views).
AEs related to the PLF grafting material or posterior fixation up to 24 months | 24 months
  A summary of AEs related to the PLF grafting material or posterior fixation up to 24 months.
Secondary surgeries related to the PLF grafting material or posterior fixation up to 24 months | 24 months
  A summary of secondary surgeries related to the PLF grafting material or posterior fixation up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chetan Patel, Principal Investigator — Spine Health Institute
Locations (17):
- United States (17):
  - University of California, Davis, Sacramento, California
  - Spine Colorado, Durango, Colorado
  - The Steadman Clinic, Vail, Colorado
  - The Spine Health Institute, Altamonte Springs, Florida
  - Foundation for Orthopedic Research and Education, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Indiana Spine Group, Carmel, Indiana
  - Fort Wayne Orthopedics, Fort Wayne, Indiana
  - The University of Kansas (KUMC), Kansas City, Kansas
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Upstate Orthopedics, East Syracuse, New York
  - New York-Presbyterian Hospital/Columbia University, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Seton Spine & Scoliosis Center, Austin, Texas
  - American Neurospine Institute PLLC, Plano, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia